CLINICAL TRIAL: NCT06210945
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Proof of Biology Study to Evaluate the Safety, Tolerability, and Activity of CM-101 in Patients With Systemic Sclerosis
Brief Title: Study to Evaluate the Safety, Tolerability, and Activity of CM-101 in Patients With Systemic Sclerosis
Acronym: ABATE
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: pending financial resources
Sponsor: ChemomAb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-101-SSC-203
Record Dates: First submitted 2023-08-22; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — streptococcal polysaccharide type III group B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CM-101 (Experimental): CM-101 will be administered
  Interventions: Drug: 10 mg/kg CM-101
- Placebo (Placebo Comparator): Placebo will be administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 10 mg/kg CM-101 — 10 mg/kg CM-101
  Arms: CM-101
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to assess the safety and tolerability of the anti-human CCL24 monoclonal antibody CM-101 in adult patients with systemic sclerosis (SSc). Approximately 45 patients at approximately 40 sites will be randomized in a 2:1 ratio to receive either 10 mg/kg CM-101 or placebo.

DETAILED DESCRIPTION:
This study will consist of a screening period, double-blind treatment period, open-label treatment period, and safety follow-up. Approximately 45 patients will be randomized in a 2:1 ratio to receive either 10 mg/kg CM-101 or placebo. The study drug or placebo, will be administered as a 60-minute intravenous (IV) infusion once every 3 weeks for a treatment coverage of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of systemic sclerosis based on the 2013 ACR-EULAR Classification Criteria for SSc with a disease duration of ≤7 years as defined by the date of onset of the first non-Raynaud's symptom. Systemic sclerosis may be of limited or diffuse type.
* A serum level of CCL24 ≥400 pg/mL at Screening
* Presence of one of the below confirming active disease at Screening:

  a. Skin involvement with mRSS ≥15 b. Presence of interstitial lung disease at Screening, evidenced by >10% involvement at HRCT (historic HRCT performed within 12 weeks of Screening may be used if the images are available to be sent to the central reader) and at least one of the following at Screening: i. C-reactive protein (CRP) ≥6 mg/L, or ii. Erythrocyte sedimentation rate (ESR) ≥28 mm/hr, or iii. Platelet count ≥(330,000/microliter), or iv. Serum level of CCL24 ≥1,000 pg/mL c. Current digital ulcer and at least one of the following at Screening: i. CRP ≥6 mg/L, or ii. ESR ≥28 mm/hr, or iii. Platelet count ≥330,000/μL), or iv. Serum level of CCL24 ≥1,000 pg/mL
* If under active immunosuppressive treatment for SSc, treatment must be stable

  ≥12 weeks before Screening with intention to continue with no change in dose from Screening through the end of study. Hydroxychloroquine (or similar antimalarial such as chloroquine) use is allowed and may be combined with up to one of the following:
  1. Methotrexate (maximum dose 25 mg/week),
  2. Azathioprine (maximum dose 200 mg/day),
  3. Mycophenolate mofetil (MMF)/mycophenolic acid (MPA) (maximum dose 2 g/dayMMF or equivalent).
* Oral corticosteroids of prednisone (or equivalent) ≤10 mg/day are allowed but not required and if present, must be stable for 30 days prior to Screening.
* If under treatment with the following, treatment must be stable for ≥8 weeks before Screening with the intention to continue with no change in dose from Screening through the end of study:

  1. Endothelin receptor antagonist, such as macitentan, bosentan, ambrisentan
  2. Phosphodiesterase type 5 inhibitors, such as sildenafil and tadalafil.
* Negative serum pregnancy test for biologically female patients of childbearing potential
* Men and women with reproductive potential are required to use a highly effective means of contraception through the course of the study

Exclusion Criteria:

1. Systemic sclerosis-like illness associated with environmental or ingested agents such as toxic rapeseed oil, vinyl chloride, or bleomycin.
2. Rheumatic autoimmune disease other than SSc, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, undifferentiated connective tissue disorder, polymyositis, dermatomyositis, eosinophilic fasciitis, primary Sjögren's syndrome, and eosinophilic myalgia syndrome when classification or diagnostic criteria for those diseases are met.
3. Systemic sclerosis with end-stage organ involvement at Screening, including:

   1. Currently or anticipating placement on an organ transplantation list, or has received an organ transplant
   2. Renal crisis within 6 months before Screening
   3. Interstitial lung disease with FVC% < 45 or requiring constant oxygen therapy. Oxygen used to aid sleep or exercise is allowed.
   4. Pulmonary hypertension requiring constant oxygen therapy or continuous intravenous treatment with prostaglandins. Oxygen used to aid sleep or exercise is allowed.
   5. Gastrointestinal dysmotility requiring total parenteral nutrition or hospitalization within 6 months before Screening.
4. Use of following treatment(s) during the study or within the times noted:

   1. Within 26 weeks prior to Screening: cyclophosphamide, rituximab
   2. Within 12 weeks prior to Screening: tocilizumab, thalidomide, cyclosporine, pirfenidone, or tyrosine kinase inhibitors (e.g., nintedanib)
   3. Within 6 weeks prior to Screening: ultraviolet (UV) phototherapy
   4. Within 30 days prior to Screening: systemic corticosteroids at doses greater than 10mg/day prednisone or equivalent
   5. Other monoclonal antibodies not listed, please consult with the Medical Monitor regarding appropriate discontinuation period
5. Anticipated to require the following treatments during the study: cell depleting therapy, chlorambucil, total lymphoid radiation, anti-thymocyte globulin, plasmapheresis, extra-corporeal photopheresis or bone marrow transplant. If prior use, consult Medical Monitor.
6. Participation in another research study of an investigational drug or device within 10 weeks of Screening or received treatment with any investigational agent within 30 days or 5 elimination half-lives (whichever is longer) of the investigational drug prior to Screening.
7. Prior exposure to CM-101
8. Any major surgery (including joint surgery) within 8 weeks prior to Screening or have surgery scheduled during the study duration.
9. Receipt of a live/attenuated vaccine within 10 days of study Screening.
10. Cancer, history of cancer or lymphoproliferative disorder within the previous 5 years (other than adequately treated nonmetastatic basal cell skin cancer or squamous cell skin cancer that has not recurred for at least 1 year prior to Screening; history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to Screening).
11. Concurrent serious medical condition which, in the opinion of the Investigator, makes the patient inappropriate for this study such as but not limited to poorly controlled chronic heart failure, clinically meaningful arrhythmia, severe pulmonary or systemic hypertension, hepatic impairment, poorly controlled diabetes, unstable atherosclerotic cardiovascular disease, or severe peripheral vascular disease.
12. Any clinically significant disease or laboratory abnormality at Screening which may interfere with the study evaluation and/or safety of the patient including the following:

    1. hemoglobin <9 g/dL
    2. absolute neutrophils <1.0 × 10-9/L
    3. white blood cells (WBC) <3,000/mm3
    4. platelets <100,000/mm3
    5. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2× upper limit of normal (ULN)
    6. total bilirubin >1.5× ULN.
13. History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV), or a previously positive result for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), or anti-HIV 1 or 2. Local testing may be performed based on Investigator judgment if there are no historical values or there is an indication for testing.
14. Known active bacterial, viral, fungal, mycobacterial, or other systemic infection including any infected ulcer(s); or any major episode of infection requiring hospitalization or treatment with IV antimicrobials within 8 weeks of Screening; or any infection requiring antibiotic therapy within 2 weeks of Screening.
15. History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies.
16. Currently pregnant or breastfeeding at entry into this study.
17. History of severe depression, psychosis, or suicidal ideation, or a history of alcohol abuse or drug addiction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by treatment-emergent adverse events (TEAEs) | 24-weeks
  Safety and tolerability will be assessed by treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
To evaluate change from Baseline in serum biological markers - growth factors and cytokines | 24 weeks
  To evaluate change from Baseline in serum biological markers, including but not limited to growth factors and cytokines (IL6, CCL2, CXCL9, CXCL10, CXCL11, and C-X3-C motif ligand [CX3CL]1).
To evaluate change from Baseline in serum biological markers - adhesion molecules | 24 weeks
  To evaluate change from Baseline in serum biological markers - adhesion molecules (intercellular adhesion molecule 1 [ICAM-1], P-selectin, vascular cell adhesion protein 1 [VCAM-1], and E-selectin).
To evaluate change from Baseline in serum biological markers - vascular | 24 weeks
  To evaluate change from Baseline in serum biological markers - vascular (vascular endothelial growth factor [VEGF], Endothelin-1, and brain natriuretic peptide [BNP])
To evaluate change from Baseline in serum biological markers - lung injury | 24 weeks
  To evaluate change from Baseline in serum biological markers - lung injury (Krebs von den Lungen 6 [KL-6]
To evaluate change from Baseline in serum biological markers - surfactant protein D | 24 weeks
  To evaluate change from Baseline in serum biological markers - surfactant protein D [SP-D], and CCL18)
To evaluate change from Baseline in serum biological markers - extracellular matrix related markers | 24 weeks
  To evaluate change from Baseline in serum biological markers - extracellular matrix related markers (collagens, matrix metalloproteinases [MMP]s, tissue inhibitors of metalloproteinases [TIMPs], and ELF).
Observed maximum plasma concentration - Cmax | 24 weeks
  To characterize the PK properties of CM-101 following repeated administrations of CM-101
Time to reach the observed maximum plasma concentration - Tmax | 24 weeks
  To characterize the PK properties of CM-101 following repeated administrations of CM-101
Area under the plasma concentration-time curve extrapolated to infinity, calculated as: AUC∞ = AUClast + Clast/λz, where AUClast is the last measurable concentration - AUC∞ | 24 weeks
  To characterize the PK properties of CM-101 following repeated administrations of CM-101
Elimination rate constant, determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve - λz | 24 weeks
  To characterize the PK properties of CM-101 following repeated administrations of CM-101
To evaluate target engagement in serum | 24 weeks
  To evaluate target engagement in serum following multiple repeated administrations of CM-101 dosing by analyzing CCL24 and CM-101 levels
anti-drug antibodies | 24 weeks
  To evaluate the development of anti-drug antibodies following repeated administrations of CM-101

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Frankel, MD, Study Director — ChemomAb Ltd.
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States